CLINICAL TRIAL: NCT02964741
Title: Investigation and Modulation of the Mu-Opioid Mechanisms in Migraine (in Vivo)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to COVID-19
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, DMedSc, Assistant Professor of Biologic and Materials Science, School of Dentistry and Research Assistant Professor, Center for Human Growth & Development, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00107286; R01NS094413 (NIH)
Record Dates: First submitted 2016-10-07; First posted 2016-11-16 (Estimated); Results first posted 2022-07-12 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-07

CONDITIONS: Migraine
Keywords: Episodic Migraine; Headache; Opioid
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Migraine Patients Active Group (Active Comparator): Episodic migraine patients will be randomized (Taves method) to receive high-definition transcranial direct current stimulation (HD-tDCS*) as 20 minute sessions, once daily for 10 days (M-F for 2 weeks).
  *Active Comparator
  Interventions: Device: Active Comparator
- Migraine Patients Sham Group (Sham Comparator): Episodic migraine patients will be randomized (Taves method) to receive high-definition transcranial direct current stimulation (HD-tDCS*) as 30-second administrations at the beginning and end of each 20 minute session, once daily for 10 days (M-F for 2 weeks).
  *Sham Comparator
  Interventions: Device: Sham Comparator
- Healthy Control Group (No Intervention): Healthy Volunteers will be asked to undergo baseline assessments only (including imaging, but no brain stimulation).
  Healthy volunteer data (n </= 10) may be used from a prior study (NINDS-K23062946 project [IRBMED #HUM00027383; Dr. Alexandre DaSilva, Principal Investigator]). Consent to use data for a future study was obtained in the informed consent document at the time of participation.

INTERVENTIONS:
Device: Active Comparator — non-invasive brain stimulation (active protocol)
  Other Names: HD-tDCS (active protocol)
  Arms: Migraine Patients Active Group
Device: Sham Comparator — non-invasive brain stimulation (sham protocol)
  Other Names: HD-tDCS (sham protocol)
  Arms: Migraine Patients Sham Group

SUMMARY:
This study investigates whether non-invasive brain stimulation, given for 20 minutes/once per day for ten days (M-F) can reduce migraine pain. Thirty patients will receive this treatment, while thirty will receive a "sham" procedure. Up to thirty healthy volunteers will be asked to undergo baseline assessments only (imaging, but no brain stimulation). Healthy volunteer data may be used from a prior study (NINDS-K23062946 project [IRBMED #HUM00027383; Dr. Alexandre DaSilva, Principal Investigator]).

DETAILED DESCRIPTION:
Migraine is a debilitating chronic condition that affects most of the patient's existence, from childhood to late adulthood. During frequent headache attacks, its sufferers show marked increased sensitivity to noxious (hyperalgesia) and even non-noxious stimuli, a phenomenon called cutaneous allodynia that affects 63% of the patients. Although MRI-based techniques have provided insights into some brain mechanisms of migraine, many questions regarding its molecular impact in the brain are still unanswered. The overall goal of this project is to provide a detailed understanding of the µ-opioid receptor mediated transmission in the brain of migraine patients, one of the most important central pain regulatory systems in humans, with the long-term objective of developing more focused neuromechanism-driven methods for migraine research and therapy.

Preliminary studies from an earlier project (NINDS-NIHK23 NS0629946) using positron emission tomography (PET) with [11C] carfentanil, a selective radiotracer for μ-opioid receptor (μOR), have indicated that there is a decrease in µOR availability (non-displaceable binding potential; BPND) in the brain of migraine patients during the headache attacks and allodynia, including areas like thalamus and periaqueductal gray matter (PAG). µOR BPND is an objective measurement, in vivo, of endogenous μ-opioid availability, and its acute reduction reflects the activation of this neurotransmitter system. This is arguably one of the neuromechanisms most centrally involved in pain regulation, affecting multiple elements of the pain experience. Moreover, MRI-based reports have found that those findings co-localize with neuroplastic changes in migraine patients. Conventional therapies are unable to selectively target those dysfunctional brain regions, and there is a paucity of data on how to reverse embedded neuroplastic molecular mechanisms when available medications and surgical therapies fail. Several studies with motor cortex stimulation (MCS) have shown that epidural electrodes in the primary motor cortex (M1) are effective in providing analgesia in patients with refractory central. The rationale for MCS stimulation is based in part on the thalamic dysfunction noticed in chronic pain and migraine, and also on studies demonstrating that MCS significantly changes thalamic activity. Evidently, the invasive nature of such a procedure limits its indication to highly severe chronic pain disorders. New non-invasive brain neuromodulatory methods for M1, such as transcranial direct current stimulation (tDCS), can now safely modulate and activate the µOR system, providing relatively lasting pain relief in chronic pain patients and migraine. However, the electric fields generated by its most conventional analgesic montage are widely spread across the brain, lacking specificity on the pain-related structures directly targeted. Recently, a novel high-definition tDCS (HD-tDCS) montage created by our group was able to reduce exclusively "contralateral" sensory-discriminative clinical pain measures (pain intensity/area) in chronic patients by targeting more precisely the putative M1 region. It is hoped that this montage will provide durable relief of pain for this episodic migraine population.

This is a phase 2, single center, two-arm, double-masked, randomized investigation and modulation of the µ-opioid mechanisms in migraine (in vivo). We will enroll 60 patients with episodic migraine (30 for the active M1 HD-tDCS group and 30 for a sham group). Each participant will undergo a sequence of events and evaluations that will include baseline assessments, 10 days of HD-tDCS, pre- and post-PET and MRI scans, and questionnaires to evaluate pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Episodic migraine (ICHD-3-beta) for at least 6 months, with at least one attack per month and less than 15 attacks per month
* No intake of opiate medication for the past six months
* No overuse of analgesic medication, defined as regular intake on ≥15 days per month for more than 3 months
* Willing to limit the introduction of new treatments for headache management

Exclusion Criteria:

* Presence of any other systemic or chronic pain disorder
* History or current evidence of a psychotic disorder (e.g. schizophrenia) or substance abuse; bipolar or severe major depression, as evidenced by Beck Depression score of ≥ 30
* History of neurological disorder (e.g. epilepsy, stroke, neuropathy, neuropathic pain)
* Prior use of tDCS
* Current use of opioid pain medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre F DaSilva, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim M, Kim DJ, Nascimento TD, DaSilva AF. High-definition tDCS over primary motor cortex modulates brain signal variability and functional connectivity in episodic migraine. Clin Neurophysiol. 2024 May;161:101-111. doi: 10.1016/j.clinph.2024.02.012. Epub 2024 Feb 15. PMID 38460220
- [Derived] DaSilva AF, Kim DJ, Lim M, Nascimento TD, Scott PJH, Smith YR, Koeppe RA, Zubieta JK, Kaciroti N. Effect of High-Definition Transcranial Direct Current Stimulation on Headache Severity and Central micro-Opioid Receptor Availability in Episodic Migraine. J Pain Res. 2023 Jul 21;16:2509-2523. doi: 10.2147/JPR.S407738. eCollection 2023. PMID 37497372

RESULTS

PARTICIPANT FLOW:
Groups:
- Migraine Patients Active Group: Episodic migraine patients will be randomized (Taves method) to receive high-definition transcranial direct current stimulation (HD-tDCS*) as 20 minute sessions, once daily for 10 days (M-F for 2 weeks).
  *Active Comparator
  Active Comparator: non-invasive brain stimulation (active protocol)
- Migraine Patients Sham Group: Episodic migraine patients will be randomized (Taves method) to receive high-definition transcranial direct current stimulation (HD-tDCS*) as 30-second administrations at the beginning and end of each 20 minute session, once daily for 10 days (M-F for 2 weeks).
  *Sham Comparator
  Sham Comparator: non-invasive brain stimulation (sham protocol)
Period: Overall Study
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group | Healthy Control Group
Started | 15 | 13 | 12
Completed | 13 | 12 | 12
Not Completed | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — claustrophobia | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group | Healthy Control Group | Total
Number analyzed (Participants) | 13 | 12 | 12 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 12 | 37
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (13.8) | 30.3 (8.8) | 32.4 (15.3) | 30.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 11 | 33
  Male | 2 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 11 | 11 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 5
  White | 9 | 9 | 7 | 25
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 12 | 37

OUTCOME MEASURES:

1. Primary Outcome: Days With Moderate-to-severe Headache
Description: Moderate to severe headache is defined by the pain over 3 in an Numeric Rating Scale (NRS) ranging from 0 to 10 between end of treatment and one month follow-up.
Time Frame: End of treatment - over 1 month follow-up
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
Number analyzed (Participants) | 13 | 12
days | 2.9 [2.1 to 3.9] | 3.3 [2.4 to 4.4]

2. Primary Outcome: Responder Rate
Description: Number of participants who showed a 50% reduction of days with moderate-to-severe headache compared to baseline.
Time Frame: End of treatment - over 1 month follow-up
Measure: Number; unit: participants
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
Number analyzed (Participants) | 13 | 12
participants | 10 | 6

3. Secondary Outcome: Change in Pain Intensity Level Measured by the Visual Analog Scale in Migraineurs (Active or Sham)
Description: Visual Analog Scale measures pain on a 0 to 10 scale, where 0 is "no pain" and 10 is "worst possible pain"
Time Frame: Approximately 45 days (Screening Visit [Original Baseline] to Follow Up #2 [28-days post-HD-tDCS treatment])
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
Number analyzed (Participants) | 13 | 12
score on scale | -4.1 [-5.3 to -2.8] | -4.4 [-5.7 to -3.1]

4. Secondary Outcome: Moderate to Severe Headache
Description: Percentage of participants having moderate-to-severe headache between end of treatment and one month follow-up.
  Defined as a response greater than 3 on the (0-10) NRS scale
Time Frame: End of treatment - over 1 month follow-up
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
Number analyzed (Participants) | 13 | 12
percentage of participants | 61.5 [35.1 to 88.0] | 66.7 [40.0 to 93.3]

5. Secondary Outcome: Use of Rescue Medication
Description: Percentage of participants who used rescue medication between end of treatment and one month follow-up
Time Frame: End of treatment - over 1 month follow-up
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
Number analyzed (Participants) | 13 | 12
percentage of participants | 38.5 [12.0 to 64.90] | 66.7 [40.0 to 93.3]

6. Secondary Outcome: Change in Mu-opioid Receptor Non-displaceable Binding Potential (BPND) in the Brains of Migraineurs During Sustained Thermal Pain Threshold Stress Challenge Subsequent to Treatment by HD-tDCS (Active or Sham).
Description: Mu-opioid receptor BPND at PET #2 will be subtracted from mu-opioid receptor BPND at PET #1.
  PET #1 occurs during the week before HD-tDCS treatment begins. PET #2 occurs during the week after the final HD-tDCS treatment is completed.
Time Frame: Time between PET #1 and PET #2 is typically 21 days (minimum 17 days; maximum 42 days).
Measure: Mean (Standard Deviation); unit: non-displaceable binding potential
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
Number analyzed (Participants) | 13 | 11
non-displaceable binding potential | 0.15 (0.09) | -0.10 (0.11)

7. Secondary Outcome: Change in Mu-opioid Receptor Non-displaceable Binding Potential (BPND) in the Brains of Migraineurs at Rest Subsequent to Treatment by HD-tDCS (Active or Sham).
Description: as for outcome 6
Time Frame: Time between PET #1 and PET #2 is typically 21 days (minimum 17 days; maximum 42 days).
Measure: Mean (Standard Deviation); unit: non-displaceable binding potential
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
Number analyzed (Participants) | 13 | 11
non-displaceable binding potential | 0.07 (0.13) | -0.15 (0.13)

ADVERSE EVENTS:
Time Frame: During the 2-weeks of HD-tDCS treatment
Description: Adverse Events were collected using a questionnaire that reflects common side effects of tDCS treatment. The questionnaire was administered before and after each of 10 tDCS treatment sessions. All of the adverse events reported were expected and mild in severity.
Arm/Group | Migraine Patients Active Group | Migraine Patients Sham Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 12/13 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migraine Patients Active Group (N=13) | Migraine Patients Sham Group (N=12)
Headache (Investigations) | 6 | 4
Neck pain (Investigations) | 6 | 3
scalp pain (Investigations) | 4 | 4
scalp burns (Investigations) | 2 | 4
tingling (Investigations) | 7 | 11
skin redness (Investigations) | 1 | 1
sleepiness (Investigations) | 8 | 8
trouble concentrating (Investigations) | 2 | 4
other (mild forms of dizziness, scalp tenderness, mild itching, etc) (Investigations) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT02964741/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT02964741/ICF_001.pdf